CLINICAL TRIAL: NCT04720560
Title: Role of Regulatory B Cells in the Pathogenesis of Metabolic Associated Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Doctor, Assiut University
Other Study IDs: MAFLD
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: regulatory B cell by flow cytometry — 4-Evaluation of the Frequency of regulatory B cells (Bregs) by Flow Cytometry Using flow cytometry, circulating Bregs will be detected using FITC-conjugated-CD38, PE-conjugated-CD24 (Bioscience, USA), and PerCP-conjugated CD19 (BD Bioscience, USA). Briefly, 100 µl of blood sample will be incubated with 10 µL of CD24, CD38 and CD19 for 20 minutes at 4 °C in the dark. Following incubation, RBCs will be lysed and washed. Cells will be fixed and permeabilized then stained with APC-conjugated IL-10 (BD Bioscience, San Jose, CA, USA) and analysis will be done by FACS Calibur flow cytometry with CellQuest software (Becton Dickinson Biosciences, San Jose, CA, USA).
  An isotype-matched negative control will be used for each sample. Forward and side scatter histograms will be used to define the lymphocytes population. CD19+ IL-10+ B cells will be gated, then the expression of CD38 and CD24 on the CD19+B cells will be detected. Bregs will be identified as CD19+ IL-10+CD24+hiCD38+hi cells.

SUMMARY:
To evaluate the role of regulatory B cells in the pathogenesis of metabolic associated fatty liver disease patients.

DETAILED DESCRIPTION:
The prevalence of non-alcoholic fatty liver disease (NAFLD) increases rapidly in recent decades. NAFLD has become a major public health problem in the whole world, and it is considered as the main cause for the chronic liver diseases (Feng, 2020).

Eslam et al. (2020) recently published an international expert consensus statement about a new definition of metabolic dysfunction-associated fatty liver disease (MAFLD) to replace non-alcoholic fatty liver disease (NAFLD).

The new nomenclature of MAFLD is based on the presence of steatosis in >5% of hepatocytes and the absence of excessive alcohol consumption or other causes of chronic liver disease, diagnosis of MAFLD could be established on the presence of hepatic steatosis in combination with one of the following three criteria: overweight/obesity; presence of type 2 diabetes mellitus; or evidence of metabolic dysregulation (Eslam et al. (2020).

Metabolic dysregulation is defined as having at least 2 of the following metabolic risk abnormalities: high waist circumference, high blood pressure, high cholesterol, pre-diabetes, insulin resistance, and high plasma C-reactive protein levels (Eslam et al. (2020).

New diagnostic criteria for MAFLD were proposed, in which hepatic steatosis (HS) detected either by imaging techniques, blood biomarkers/scores or by liver histology (Bedogni et al., 2006; Wong et al., 2019).

On the other hand, NAFLD is commonly associated with one or more component of metabolic syndrome such as obesity, diabetes mellitus, and dyslipidemia and is defined as the presence of ≥ 5% hepatic steatosis in histological examination without evidence of hepatocellular injury such as hepatocyte ballooning (Chalasani et al., 2018).

Around 20% of patients with NAFLD develop non-alcoholic steatohepatitis (NASH) which may progress to cirrhosis, however the most common cause of death in NAFLD patients is cardiovascular disease, and NAFLD is the third most common cause of hepatocellular carcinoma (Matteoni et al., 1999; Chalasani et al., 2018).

The spectrum of NAFLD ranges from simple fatty liver with little inflammation to non-alcoholic steatohepatitis (NASH) with liver inflammation and fibrosis. The global prevalence of NAFLD is about 25.2% whereas the limited number of studies from Africa reports 13% (Younossi et al., 2016).

"Burned out" NAFLD can be a hidden cause of cryptogenic cirrhosis. So, early diagnosis, and treatment of NAFLD and underlying predisposing factors are important to avoid liver damage which may progress to liver cell failure (Paul, 2020).

NAFLD is strongly associated with MS and is currently considered as the hepatic manifestation of MS. In addition, obesity is a common risk factor for NAFLD (fan et al., 2008; Chen et al., 2011; Medina-Santillán et al., 2013).

Liver is not only the largest metabolic organ, but also it act as an immunological organ. Immune cells including liver resident macrophages )Kupffer cells, KCs( and lymphocytes account for 10-20% of total cells in the liver (Racanelli et al., 2006; Gao et al., 2008).

These immune cells cross the blood from gastrointestinal tract, which contains abundant antigens from outside and sometime pathogens under pathological conditions, to maintain a unique immune tolerance microenvironment (Racanelli et al., 2006).

However, when excessive fat deposited in the hepatocytes and metabolic status was changed, the immune microenvironment was found to be also changed. Numerous studies indicated that different immune cells in the liver (both innate and adaptive) played critical roles in the pathogenesis of NAFLD and NASH(Feng, 2020).

Innate immune system includes KCs/infiltrated macrophages, neutrophils, dendritic cells (DCs), natural killer (NK) cells, while adaptive immune system includes conventional T cells, natural killer T (NKT) cells and B cells(Feng, 2020).

Smith et al. (2003) examined healthy human donor livers and detected the B cells located in the portal tracts and those scattered throughout the liver.

B cells are specialized adaptive immune cells producing antibodies, it can also secrete cytokines and regulate the activation and function of other cells. Little studies focused on the role of B cells in the pathogenesis of NAFLD, especially direct effects. One study showed that increased production of T-helper 1 cell (Th1) cytokines, such as IL-6 and TNF-a, which were found in intrahepatic B cells in mice fed with high-fat diet. These cytokines may promote Th1 cell differentiation and contribute to inflammation in NAFLD (Zhang et al., 2016).

As regard role of B cells in the pathogenesis of metabolic syndrome (MS) which promote inflammation in obesity and type 2 diabetes mellitus (T2DM) through modulation of T-cell function and an inflammatory cytokine profile and they also promote insulin resistance (IR) through the production of pathogenic IgG2a. Meanwhile, B cells can regulate T cells via a major histocompatibility complex-dependent manner and promote inflammation mediated by T cells in both obese mice and T2DM patients (Jagannathan et al., 2009; Winer et al., 2011; DeFuria et al., 2013).

NAFLD is strongly associated with MS and is currently considered as the hepatic manifestation of MS. In addition, obesity is a common risk factor for NAFLD (fan et al., 2008; Chen et al., 2011; Medina-Santillán et al., 2013).

Surprisingly, IgA, which is mainly produced by B cells, has been reported to be positively related to the stages of fibrosis in patients with NAFLD. The B cell activating factor (BAFF), which regulates the development and maturation of B cells, was found to be increased in the serum of patients with non-alcoholic steatohepatitis (NASH). All these results indicate that there are systemic changes in B cells in patients with NAFLD (Kim et al., 2009; Miyake et al., 2013; McPherson et al., 2014).

Based on the changes in humoral factors in NAFLD and the roles of B cells in MS, we hypothesized that B cells might participate in the pathogenesis of NAFLD. So, our study aimed to focus on B cells, to investigate its general changes and their functions in the pathogenesis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years old and was diagnosed as fatty liver based on clinical examination, laboratory investigations and imaging techniques.

Exclusion Criteria:

* 1-Patients aged ≤18 years old. 2-Pregnancy. 3-Presence of malignancy. 4-Type I DM. 5-Fatty liver patients on treatment by statin derivatives or other medications. 6- Fatty liver patients undergone bariatric surgeries.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. After obtaining the appropriate consents, data pertaining to clinical history (name, age, sex, residence, occupation, co-morbidities… diabetes, hyperlipidemia, hypertension, ischemic heart disease, special habits; such as alcohol intake).
  2. Imaging techniques, such as ultrasonography (US), fibroscan with CAP and/or computed topography (CT) and /or MRI.
  3. Blood samples will be collected for liver function tests, lipid profile and CRP.
  4. Evaluation of the Frequency of regulatory B cells (Bregs) by Flow Cytometry
  5. Six measurements will be obtained (sex, age, height, weight, body mass index, and abdominal girth, waist circumference).
  Calculation of fatty liver index, (FLI) will be done. The fatty liver index (FLI), is an algorithm based on waist circumference, body mass index (BMI), triglyceride, and gamma-glutamyl-transferase (GGT).
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Role of regulatory B cells in the pathogenesis of metabolic associated fatty liver disease | baseline
  To evaluate the role of regulatory B cells in the pathogenesis of metabolic associated fatty liver disease patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Asyut, Egypt

REFERENCES:
- [Background] Vilar-Gomez E, Chalasani N. Non-invasive assessment of non-alcoholic fatty liver disease: Clinical prediction rules and blood-based biomarkers. J Hepatol. 2018 Feb;68(2):305-315. doi: 10.1016/j.jhep.2017.11.013. Epub 2017 Dec 2. PMID 29154965